CLINICAL TRIAL: NCT03913013
Title: Technology-Enhanced Family-Focused Treatment for Adolescents at High Risk for Mood Disorders
Brief Title: Technology Enhanced Family Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#18-000906; R34MH117200 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Mood Disorders; Bipolar Disorder; Major Depression
Keywords: Family Therapy
MeSH Terms: conditions — Mood Disorders; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The investigation is comparing youth who receive family-focused treatment with the MyCoachConnect (FFT-MCC) mobile application (assessments, skill training, psychoeducation) to youth who receive FFT plus only the assessment components of the MCC app (FFT-Assess) on symptomatic outcome and family functioning over 27 weeks.
Who Masked: Outcomes Assessor
Masking Description: The Outcomes assessor will be unaware of whether the patient is in FFT-MCC or FFT-Assess.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFT with MCC App (FFT-MCC) (Experimental): Youth in this study arm will receive 12 sessions of FFT (psychoeducation, communication skills training, and problem-solving skills training) with their parents and siblings. They and their parents will make regular mobile app ratings of mood, sleep, family functioning, stress, and perceived criticism. Children and parents will call into a voice-activated phone system and be asked to speak freely for 3-5 minutes about their health and family functioning. They will be guided through 12 lesson plans in which they practice skills such as active listening or identifying prodromal signs of episodes, paralleling what they are learning in sessions. The clinician will be able to set a weekly skill training assignment and observe the family's practice of the skill between sessions. They will adapt session content accordingly.
  Interventions: Behavioral: Family-Focused Treatment with MCC App
- FFT with App Assessments only (FFT-Assess) (Active Comparator): Youth in this condition will receive the same 12 sessions of FFT, but the app will be limited to daily and weekly assessments of their mood, sleep, stress, and family functioning. The app will not provide the skill training offered in the FFT-MCC condition.
  Interventions: Behavioral: Family-Focused Treatment with MCC App

INTERVENTIONS:
Behavioral: Family-Focused Treatment with MCC App — 12 sessions of family-focused therapy plus use of a mobile app that enhances the skill training taught in the sessions.

SUMMARY:
The investigators propose to enhance the scalability of family-focused therapy (FFT), a 12-session evidence-based therapy for youth at high risk for mood disorders, through augmentation with a novel mobile phone application called MyCoachConnect (MCC). In adolescents with mood instability who have a parent with bipolar or major depressive disorder, clinicians in community clinics will conduct FFT sessions (consisting of psychoeducation and family skills training) supplemented by weekly MCC "real time" assessments of moods and family relationships; based on results of these assessments and the family's progress in treatment, clinicians will then push personalized informational and coaching alerts regarding the practice of communication and problem-solving skills. The investigators hypothesize that the augmented version of FFT (FFT-MCC) will be more effective than FFT without coaching/informational alerts in altering treatment targets and in stabilizing youths' mood symptoms and quality of life.

DETAILED DESCRIPTION:
The investigative group has shown in several randomized trials that family-focused therapy (FFT) for symptomatic youth at high-risk for bipolar disorder - consisting of psychoeducation and family communication and problem solving skills training - is an effective adjunct to pharmacotherapy in hastening symptomatic recovery. However, between 50%-60% of high-risk youth still have residual mood symptoms and functional impairment after 18 weeks of FFT. In prior studies, two constructs have emerged as predictors of lack of response to treatment: mood instability in the child and expressed emotion (EE) in parents (i.e., frequent critical comments or hostility). In adolescents (ages 12-18) with a parent with bipolar disorder or major depressive disorder, the investigators hypothesize that augmenting FFT with frequent and targeted interventions in the home setting through a Smartphone app (MyCoachConnect, or MCC) will (a) have a greater and more rapid impact than standard FFT on the targeted mechanisms of mood instability in adolescents and EE in parents, and (b) as a result, enhance symptom resolution and functioning in adolescents. To be eligible, adolescents must score high on parent-rated measures of mood instability, and have at least one parent who is high-EE by speech sample coding criteria. The MCC app will record weekly open speech samples from parents and children and daily and weekly mood ratings from adolescents. The app assessments will be fed back to the FFT clinician, who will use this information to "push" recommendations for mood regulation, communication, and problem-solving strategies (linked to the FFT modules) for parents and youth. In year 1, the investigators will conduct an open trial (n=25) to determine (a) the feasibility and acceptability of FFT with mobile coaching (FFT-MCC), as given by clinicians in community settings, and (b) associations between online/speech feature proxies of the targets (mood instability and EE as measured weekly by MCC) and standard measures of the targets. In years 2 and 3 the investigators will conduct a 60-case randomized clinical trial in which families are assigned to FFT with MCC skills coaching or FFT with MCC assessments only, with no skills coaching. The primary hypotheses are that FFT-MCC will be acceptable to parents, adolescents and clinicians, and more effective than FFT without MCC coaching in engaging the targets of mood instability and EE and promoting improvements in adolescents' mood symptoms and quality of life over 27 weeks. The study will facilitate the translation of a technological augmentation to an evidence-based family intervention, with the goal of increasing treatment access among families with mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and has access to smart-phones, a tablet, or computer
* Age 13-19 years old
* One parent with diagnosis of bipolar disorder type I, bipolar disorder type II, or
* major depressive disorder.
* At least one parent is rated high in perceived criticism of the child.
* Child shows evidence of mood instability
* Child is not currently in individual therapy.

Exclusion Criteria:

* Over 6 on the Autism Spectrum Disorder screener
* a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition manic episode of bipolar I disorder has occurred in the past 2 weeks
* history of persistent psychotic symptoms that have not remitted when mood states remit.
* intelligence quotient below 70 from school records
* Any significant and persistent substance or alcohol abuse in the prior 3 months
* Previously received a full course (i.e., 10-12 sessions) of FFT
* Current, active sexual abuse, physical abuse, or domestic violence.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armen Arevian, MD, Principal Investigator — University of California, Los Angeles; David J Miklowitz, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Child and Adolescent Mood Disorders Program, UCLA School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will submit digital files to the NIH Freedom of Information Office Coordinator containing all raw data, variable coding information, and copies of measures. The investigators will share the data with other investigators through the National Database for Clinical Trials Related to Mental Illness.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One year following completion of the trial.
Access Criteria: Meta-analyses

REFERENCES:
- [Background] Miklowitz DJ, Chung B. Family-Focused Therapy for Bipolar Disorder: Reflections on 30 Years of Research. Fam Process. 2016 Sep;55(3):483-99. doi: 10.1111/famp.12237. Epub 2016 Jul 29. PMID 27471058
- [Derived] Miklowitz DJ, Weintraub MJ, Denenny DM, Merranko JA, Hooley JM. Parental expressed emotion, family conflict, and symptom severity in adolescent offspring of parents with mood disorders. J Affect Disord. 2025 Nov 15;389:119620. doi: 10.1016/j.jad.2025.119620. Epub 2025 Jun 9. PMID 40494497
- [Derived] Miklowitz DJ, Ichinose MC, Weintraub MJ, Merranko JA, Singh MK. Family Conflict, Perceived Criticism, and Aggression in Symptomatic Offspring of Parents With Mood Disorders: Results From a Clinical Trial of Family-Focused Therapy. JAACAP Open. 2024 Feb 28;3(1):73-84. doi: 10.1016/j.jaacop.2024.01.008. eCollection 2025 Mar. PMID 40109484
- [Derived] Miklowitz DJ, Weintraub MJ, Ichinose MC, Denenny DM, Walshaw PD, Wilkerson CA, Frey SJ, Morgan-Fleming GM, Brown RD, Merranko JA, Arevian AC. A Randomized Clinical Trial of Technology-Enhanced Family-Focused Therapy for Youth in the Early Stages of Mood Disorders. JAACAP Open. 2023 Sep;1(2):93-104. doi: 10.1016/j.jaacop.2023.04.002. Epub 2023 Apr 26. PMID 38094620
- [Derived] Miklowitz DJ, Weintraub MJ, Posta F, Walshaw PD, Frey SJ, Morgan-Fleming GM, Wilkerson CA, Denenny DM, Arevian AA. Development and Open Trial of a Technology-Enhanced Family Intervention for Adolescents at Risk for Mood Disorders. J Affect Disord. 2021 Feb 15;281:438-446. doi: 10.1016/j.jad.2020.12.012. Epub 2020 Dec 8. PMID 33360365
- See also: UCLA Child and Adolescent Mood Disorders program — https://www.semel.ucla.edu/champ

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant enrollment numbers reflect youth participants enrolled.
Period: Overall Study
Arm/Group | FFT With MCC App (FFT-MCC) | FFT With App Assessments Only (FFT-Assess)
Started | 32 | 33
Completed | 29 | 30
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FFT With MCC App (FFT-MCC) | FFT With App Assessments Only (FFT-Assess) | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age, Mean yrs (SD) | 15.6 (1.7) | 15.9 (1.5) | 15.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 26 | 21 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 3 | 3
  White | 23 | 23 | 46
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Diagnosis [Count of Participants; unit: Participants]
  Depressive spectrum disorder | 26 | 27 | 53
  Bipolar spectrum disorder | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Average Depression Symptom Scores Over 27 Weeks on the Adolescent Longitudinal Interval Follow-up Evaluation
Description: Adolescent Longitudinal Interval Followup Evaluation (ALIFE), a measure of weekly depressive symptom fluctuation based on an interview with the child and parent (or parent unit). The primary outcome variable for this study is the average of the ALIFE weekly consensus ratings. For the ALIFE, an independent evaluator rates the child's level of depression each week for 27 weeks on a Psychiatric Status Rating (PSR) scale ranging from 1 (asymptomatic) to 6 (extremely symptomatic). Scores of 5 or higher are considered full syndromal (e.g., for major depressive disorder) and scores of 1-2 are considered remitted. For each of 27 weeks the evaluator provides a separate rating based on the child interview and parent interview and then calculates a weekly consensus rating per ALIFE developer guidelines.
Time Frame: 27 weeks (average rating across this time period)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FFT With MCC App (FFT-MCC) | FFT With App Assessments Only (FFT-Assess)
Number analyzed (Participants) | 29 | 28
score on a scale | 3.39 (1.15) | 3.09 (0.91)

2. Secondary Outcome: Mood Instability, as Rated by Parents and Children Using the Children's Affective Lability Scale (CALS)
Description: Children's Affective Lability Scale (CALS) is a 20-item parent-report survey that measures youth difficulty with affective regulation. Each item corresponds to a particular problem in affective regulation, with responses offered on a five-point scale ranging from 0 = Never or rarely occurs to 4 = 1 or more times a day). The total possible score is a sum of item scores and ranges from 0 to 80. Lower scores indicate less affective lability. In this study, a score of 20 or higher was used to indicate high mood instability.
Time Frame: Outcomes scores at 27 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FFT With MCC App (FFT-MCC) | FFT With App Assessments Only (FFT-Assess)
Number analyzed (Participants) | 28 | 28
score on a scale | 38.43 (14.12) | 33.79 (11.9)

3. Secondary Outcome: Expressed Emotion in Parents From the Five Minute Speech Sample
Description: Parental expressed emotion is a measure of critical comments, hostility, or emotional overinvolvement. The primary instrument in this study is the Five Minute Speech Sample, which is scored by an independent evaluator on number of criticisms, presence/absence of hostility, or over-involvement. One critical comment or a rating of present for hostility or over-involvement means the parent is rated high in expressed emotion, and low expressed emotion otherwise.
Time Frame: Count of participants with primary parent rated high in expressed emotion at 27 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | FFT With MCC App (FFT-MCC) | FFT With App Assessments Only (FFT-Assess)
Number analyzed (Participants) | 29 | 27
Participants | 17 | 16

4. Secondary Outcome: Free Speech Samples Coded Using the Linguistic Inquiry Word Count System.
Description: Callers are asked to speak for 3-5 minutes about how they are doing and whether anything has gone well or whether they have had difficulties. The samples will be transcribed and coded via the Linguistic Inquiry Word Count. The goal is to measure whether mood instability and expressed emotion can be captured from weekly free speech call-ins by parents or youth.
Time Frame: weekly call-ins, with linguistic counts of negative or positive words tabulated each week for 27 weeks.
Reporting Status: Not Posted

5. Secondary Outcome: Children's Global Assessment of Functioning
Description: The Children's Global Assessment of Functioning is a 1-100 rating of level of psychosocial functioning in the past 2 weeks. Higher scores indicate better functioning.
Time Frame: Means are reported at 27 weeks (study endpoint)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FFT With MCC App (FFT-MCC) | FFT With App Assessments Only (FFT-Assess)
Number analyzed (Participants) | 32 | 33
score on a scale | 65.97 (2.51) | 62.16 (2.51)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were recorded by the treating clinician and the independent evaluator at baseline, 9, 18, and 27 weeks. An Adverse Events recording form was used.
Arm/Group | FFT With MCC App (FFT-MCC) | FFT With App Assessments Only (FFT-Assess)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 5/32 | 3/33
Other Adverse Events (participants affected / at risk) | 7/32 | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FFT With MCC App (FFT-MCC) (N=32) | FFT With App Assessments Only (FFT-Assess) (N=33)
Inpatient hospitalization or Emergency Room visit (Psychiatric disorders) | 5 (5) | 3 (3) — Admission is due to psychiatric reasons- suicidal ideation or plans, psychotic symptoms
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FFT With MCC App (FFT-MCC) (N=32) | FFT With App Assessments Only (FFT-Assess) (N=33)
Self-harm, with or without suicidal ideation (Psychiatric disorders) | 7 (9) | 9 (9)

LIMITATIONS AND CAVEATS:
This study illustrates some of the limitations of mobile health interventions for youth with mood disorders. During treatment not all participants completed the weekly app check-ins or utilized the app even when encouraged to do so and provided push reminders. The present study could not evaluate the impact on clinical outcomes of adding mobile apps to standard FFT without a third group of youth who received standard FFT without any app as the comparative condition used an app for surveys.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03913013/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT03913013/SAP_001.pdf